CLINICAL TRIAL: NCT05649930
Title: Effect of Functional Power Training on Muscle Morphology and Strength of the Medial Gastrocnemius in Children With Spastic Paresis
Brief Title: Effect of Functional Power Training on Calf Muscle Length and Strength in Children With Spastic Paresis
Acronym: MegaMuscle
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Reade Rheumatology Research Institute (Other); University Ghent (Other)
Responsible Party: Principal Investigator, Babette Mooijekind, Coordinating Investigator, Amsterdam UMC, location VUmc
Other Study IDs: MegaMuscle; 2021015 (Other Grant/Funding Number: Phelps stichting voor spastici); 20210088 (Other Grant/Funding Number: JKF/KFA); AMS-2021-Innovatiecall-P5 (Other Grant/Funding Number: Amsterdam Movement Sciences)
Record Dates: First submitted 2022-11-07; First posted 2022-12-14 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Medial gastrocnemius morphology; 3D ultrasonography; Functional power training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spastic paresis: Children with spastic paresis
  Interventions: Other: Functional power training

INTERVENTIONS:
Other: Functional power training — The training consists of weighted running and walking exercises performed at high-velocity and is given three times a week for 12 weeks.

SUMMARY:
Spastic paresis (SP) is a common motor condition in children and is often caused by cerebral palsy. Skeletal muscles develop differently in children with SP due to brain damage in early development; muscle strength and muscle length are reduced compared to typically developing (TD) children. Especially, the calf muscles are affected, which particularly affects their ability to walk and to run, hindering participation in society. There are several treatments aimed to increase the range of motion of the joint by lengthening the muscle, for example botulinum toxin injections. However, these treatments can have a weakening effect on the muscle due to deconditioning from immobilization and due to paralysis.

In rehabilitation centers in the Netherlands functional power training (MegaPower) is offered to children with SP who want to walk and run better. It has been shown that this training improves calf muscle strength and performance during functional walking tests. However, the effect of MegaPower training on muscle morphology (i.a. muscle volume and length) is still unknown. Therefore, the aim of this study is to assess the effect of MegaPower training on the muscle morphology of the medial gastrocnemius in children with SP using 3D ultrasonography. It is expected that MegaPower training results in an increase of muscle volume as well as elongation of the muscle belly. Muscle volume could increase due to hypertrophy of the muscle fibers induced by the training, which could elongate the muscle belly length due to the pennate structure of the medial gastrocnemius. A double-baseline design will be applied for this study with three different measurement times (T0-T1-T2) to compare the training period (12 weeks) with a period (12 weeks) of usual care.

ELIGIBILITY:
Inclusion Criteria:

* Gross Motor Function Classification System I-III
* Children should be able to lie on their stomach for min. one minute
* Children should be able to follow instructions.

Exclusion Criteria:

* Received (one of) the following interventions within six months:
* Casting
* Botulinum toxin type-A injections
* Orthopedic surgery.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The children will be recruited from rehabilitations centres in the Netherlands.
Sampling Method: Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Muscle volume in dm^3 | 12 weeks before start training (week -12)
Muscle volume in dm^3 | At the start of training (week 0)
Muscle volume in dm^3 | At the end of the training (week 12)
Muscle belly length in mm | 12 weeks before start training (week -12)
Muscle belly length in mm | At the start of training (week 0)
Muscle belly length in mm | At the end of the training (week 12)
Tendon length in mm | 12 weeks before start training (week -12)
Tendon length in mm | At the start of training (week 0)
Tendon length in mm | At the end of the training (week 12)
Fascicle length in mm | 12 weeks before start training (week -12)
Fascicle length in mm | At the start of training (week 0)
Fascicle length in mm | At the end of the training (week 12)

SECONDARY OUTCOMES:
Isometric muscle strength of the medial gastrocnemius | At the start of training (week 0)
  Measured with a hand-held dynamometer in Nm.
Isometric muscle strength of the medial gastrocnemius | At the end of the training (week 12)
  Measured with a hand-held dynamometer in Nm.
Dynamic muscle strength | At the start of training (week 0)
  Standing heel-rise test on one leg. Measured in amount of repetitions.
Dynamic muscle strength | At the end of the training (week 12)
  Standing heel-rise test on one leg. Measured in amount of repetitions.
Functional Strength Measure (FSM) | At the start of training (week 0)
  Measurement for lower and upper limb functionality.
Functional Strength Measure (FSM) | At the end of the training (week 12)
  Measurement for lower and upper limb functionality.
1-minute-walk-test | At the start of training (week 0)
  Distance (m) covered in 1 min walking.
1-minute-walk-test | At the end of the training (week 12)
  Distance (m) covered in 1 min walking.
10m Shuttle run test | At the start of training (week 0)
  Measured in amount of steps reached.
10m Shuttle run test | At the end of the training (week 12)
  Measured in amount of steps reached.
6x15m sprint | At the start of training (week 0)
  Measured as average time (s) over 6x15 m sprint.
6x15m sprint | At the end of the training (week 12)
  Measured as average time (s) over 6x15 m sprint.
Ankle range of motion | At the start of training (week 0)
  Maximal dorsiflexion in degrees manually measured with a goniometer.
Ankle range of motion | At the end of the training (week 12)
  Maximal dorsiflexion in degrees manually measured with a goniometer.
Body weight in kg | 12 weeks before start training (week -12)
Body weight in kg | At the start of training (week 0)
Body weight in kg | At the end of the training (week 12)
Body length in m | 12 weeks before start training (week -12)
Body length in m | At the start of training (week 0)
Body length in m | At the end of the training (week 12)
Lower leg length in mm | 12 weeks before start training (week -12)
  Measured from the lateral malleolus and tibial plateau.
Lower leg length in mm | At the start of training (week 0)
  Measured from the lateral malleolus and tibial plateau.
Lower leg length in mm | At the end of the training (week 12)
  Measured from the lateral malleolus and tibial plateau.

OTHER OUTCOMES:
Medical file information | 12 weeks before start training (week -12)
  Age, gender, GMFCS-level, medical history

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein M van der Krogt, Dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Reade, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No